CLINICAL TRIAL: NCT01458184
Title: A Randomized Trial of the PhoneCare System to Improve Ambulatory Care for Patients With Chronic Diseases
Brief Title: Study of PhoneCare System to Treat Patients With Chronic Diseases
Acronym: ComplexPt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-27747
Record Dates: First submitted 2011-06-29; First posted 2011-10-24 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Disease
Keywords: risk factors for complications; precarious medical situations
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PhoneCare system (Experimental): This arm is evaluating whether utilizing the PhoneCare system aids participants with their complex health care needs.
  Interventions: Behavioral: PhoneCare system
- Control Group: without PhoneCare System (No Intervention): Subjects in this arm will receive the usual care. Usual care is defined as receiving regular care from their physicians and no additional care or intervention from the study.

INTERVENTIONS:
Behavioral: PhoneCare system — The aim of this study is to assess the effectiveness of Telephone-Linked Care for Complex Patients (TLC-C) in the care of patients with complex health care needs. TLC-C uses conversational computer telephony to monitor patients' multiple diseases between their ambulatory care visits. The system monitors patients through "virtual visits" and detects and notifies clinicians about important clinical problems to attend to. It also promotes patient self-care (e.g., medication adherence and appointment preparation).
  Other Names: TLC-C
  Arms: PhoneCare system

SUMMARY:
The aim of this study is to assess the effectiveness of Telephone-Linked Care for Complex Patients (TLC-C) in the care of patients with complex health care needs. These are patients frequently transitioning from inpatient to ambulatory care with multiple chronic diseases that tend to lead to increased health-care utilization and other socio-economic vulnerabilities. The objective is to reduce preventable hospital utilization, improve quality of life, increase satisfaction with ambulatory care, improve disease-specific metrics, and reduce net payer costs.

DETAILED DESCRIPTION:
TLC-C is a modification of an existing TLC-Multi-Disease system that targets patients with multiple chronic diseases combined with a post-hospital discharge intervention (TLC-RED-Lit). TLC-C uses conversational computer telephony to monitor patients' multiple diseases between their ambulatory care visits. The system works in both routine (patient stable) and exacerbation (patient unstable) modes. The system monitors patients through "virtual visits" and detects and notifies clinicians about important clinical problems to attend to. It also promotes patient self-care (e.g., medication adherence and appointment preparation). In emergent situations the system recommends going to the local Emergency Department (ED). In urgent situations, an alert is sent to the clinician or to his/her coverage provider. Exacerbation mode is used when the patient is discharged from a hospital inpatient service or ED or has worsening symptoms. It concentrates on the exacerbating disease and monitors patient status (improved, stable or deteriorating). Daily contact is maintained until the patient's status improves. Routine mode occurs with the patient at their baseline status and monitors the disease and the patients' self-care behaviors.

The investigators propose to perform a multi-method evaluation study of the patients, the providers, and the practice. This includes a 2-arm randomized clinical trial of TLC-C versus usual care for patients with two or more chronic diseases, at least one previous episode of acute hospital utilization over the last 12 months, and who had been recently discharged from an urban hospital. The randomized clinical trial (RCT) will evaluate the system in 440 patients followed for 6 months.

The primary outcome is acute hospital care utilization (unplanned hospitalizations and ED visits). Secondary outcomes include patient quality of life (EuroQol 5D [EQ-5D]), satisfaction (Clinician and Group Survey [G-CAHPS]), ambulatory appointment show rate and net payer costs. The investigators will explore disease specific metrics (e.g., hemoglobin A1c [HbA1c] or blood pressure). The investigators will perform formative and summative qualitative studies of the implementation of the system, its use and performance over time, and its impact on the patients, providers and the practice as a whole.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or more
* on one of Boston Medical Center (BMC)'s general medical services with an unscheduled hospitalization
* has a primary care provider in the BMC General Internal Medicine (GIM) practice or Family Medicine practice or is willing to be assigned a primary care physician (PCP) at BMC GIM or Family Medicine practice upon discharge
* once discharged, patient is planning to continue his/her primary care at BMC for the next 6 months
* communicates in English adequately to participate

Exclusion Criteria:

* patients who are admitted from hospice, nursing home or another institutional setting
* patients who are in police custody or have a suicide sitter
* patients who cannot use a telephone unassisted or who do not have regular access to either a land line or cellular telephone for the next 6 months
* patients unwilling to accept calls to his/her phone for the next 6 months
* patients currently enrolled in this study or in the RED-Lit trial
* patients unable to independently consent to participate
* patients who have sickle cell anemia
* patients responding positively to the question on the Patient Health Questionnaire (PHQ-9) regarding suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2008-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Acute Hospital Care Utilization | 3 months
Acute Hospital Care Utilization | 6 months

SECONDARY OUTCOMES:
Patient Quality of Life | 3 months
Ambulatory Appointment Show Rate | 3 months
Patient Quality of Life | 6 months
Patient Satisfaction | 6 months
  A validated, in-house designed questionnaire will be administered to subjects to assess their satisfaction with the TLC system.
Ambulatory Appointment Show Rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jack, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Marcantonio ER, McKean S, Goldfinger M, Kleefield S, Yurkofsky M, Brennan TA. Factors associated with unplanned hospital readmission among patients 65 years of age and older in a Medicare managed care plan. Am J Med. 1999 Jul;107(1):13-7. doi: 10.1016/s0002-9343(99)00159-x. PMID 10403347
- [Background] Wolff JL, Starfield B, Anderson G. Prevalence, expenditures, and complications of multiple chronic conditions in the elderly. Arch Intern Med. 2002 Nov 11;162(20):2269-76. doi: 10.1001/archinte.162.20.2269. PMID 12418941
- [Background] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354
- [Background] Stewart S, Marley JE, Horowitz JD. Effects of a multidisciplinary, home-based intervention on unplanned readmissions and survival among patients with chronic congestive heart failure: a randomised controlled study. Lancet. 1999 Sep 25;354(9184):1077-83. doi: 10.1016/s0140-6736(99)03428-5. PMID 10509499
- [Background] Dudas V, Bookwalter T, Kerr KM, Pantilat SZ. The impact of follow-up telephone calls to patients after hospitalization. Am J Med. 2001 Dec 21;111(9B):26S-30S. doi: 10.1016/s0002-9343(01)00966-4. PMID 11790365
- [Background] Friedman RH, Kazis LE, Jette A, Smith MB, Stollerman J, Torgerson J, Carey K. A telecommunications system for monitoring and counseling patients with hypertension. Impact on medication adherence and blood pressure control. Am J Hypertens. 1996 Apr;9(4 Pt 1):285-92. doi: 10.1016/0895-7061(95)00353-3. PMID 8722429
- [Background] Friedman RH, Stollerman JE, Mahoney DM, Rozenblyum L. The virtual visit: using telecommunications technology to take care of patients. J Am Med Inform Assoc. 1997 Nov-Dec;4(6):413-25. doi: 10.1136/jamia.1997.0040413. PMID 9391929
- [Background] Friedman RH, Stollerman J, Rozenblyum L, Belfer D, Selim A, Mahoney D, Steinbach S. A telecommunications system to manage patients with chronic disease. Stud Health Technol Inform. 1998;52 Pt 2:1330-4. PMID 10384677
- [Background] Friedman RH. Automated telephone conversations to assess health behavior and deliver behavioral interventions. J Med Syst. 1998 Apr;22(2):95-102. doi: 10.1023/a:1022695119046. PMID 9571516